CLINICAL TRIAL: NCT04997200
Title: Effect of Sleep Deprivation on Breathlessness and Exercise Capacity in COPD: a Randomized Crossover Trial
Brief Title: Effect of Sleep Deprivation on Breathlessness and Exercise Capacity in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Blekinge County Council Hospital (Other)
Responsible Party: Principal Investigator, Magnus Ekström, MD, PhD, Associate professor, Skane University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Version 1
Record Dates: First submitted 2021-07-21; First posted 2021-08-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: COPD
Keywords: Dyspnea; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory

STUDY DESIGN:
Intervention Model Description: Performed in randomized order on two separate days, at least seven days apart and no more than six weeks apart.
  * Intervention: A night without sleep. No daytime sleeping the day before the test. Participants are observed by staff at the trial unit during the night before the test.
  * Control: Normal night's sleep (at least six hours of sleep) in the patient's home.
  The participants wear an actigraph during 48 hours before the test to ensure adherence to the allocated condition (sleep deprivation or control).
Masking Description: The analyst analyzing the data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: One night's sleeplessness (Experimental): A night without sleep. No daytime sleeping the day before the test. Participants are observed by staff at the trial unit during the night before the test.
  Interventions: Behavioral: One night's sleeplessness
- Control: One night's normal sleep (No Intervention): A normal night's sleep (at least six hours) in the patient's home.

INTERVENTIONS:
Behavioral: One night's sleeplessness — A night without sleep. No daytime sleeping the day before the test. Participants are observed by staff at the trial unit during the night before the test.
  Arms: Intervention: One night's sleeplessness

SUMMARY:
This is a randomized controlled cross-over trial designed to measure the effect of one night's sleep deprivation on exercise endurance, ventilation and breathlessness in outpatients with COPD.

DETAILED DESCRIPTION:
Background:

Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and mortality in the world. Breathlessness and exercise limitation are cardinal symptoms in COPD with grave consequences for the patient. Even with optimal COPD treatment a large number of these patients experience a breathlessness which limits their everyday life. Physical activity is the main trigger of breathlessness in daily life, but knowledge is limited on how other factors may affect exercise performance, breathing and exertional breathlessness in patients with COPD.

Sleep deprivation is common in the population in patients with COPD, and especially in patients with worsening health status and during hospitalizations. As many as 40-45% of patients older than 70 experience sleep deprivation during hospitalization. As many as 21 % of patients with COPD have a disturbed sleep. A recent study on healthy young males who breathed against an inspiratory resistance showed that one night's sleep deprivation significantly reduced their respiratory endurance and induced worse and more disturbing breathlessness.

Little is known how sleep loss affects patients with COPD in an outpatient setting. Several studies have evaluated the effect of sleep deprivation on exercise capacity in young healthy adults. However, very few studies have examined the effect of sleep deprivation on the exercise capacity or exertional breathlessness in patients with COPD; most data pertain to observational studies where no intervention took place and data from a randomized controlled trial (RCT) is needed. The presence of disturbed sleep in patients with COPD - and especially in relation to worsenings and hospitalizations, could have a marked detrimental effect on their breathing, increase suffering from distressing breathlessness and potentially increase the risk of adverse health outcomes and worse prognosis. Directed actions to improve sleeping in these settings could in that case improve the patients' outcomes.

Aim:

To test the effect of one sleepless night on breathlessness, exercise endurance and ventilation in patients with COPD.

Method:

This is a randomized (ratio 1:1), controlled, crossover trial of the effect of one night's sleep deprivation vs. normal sleep on exercise endurance, ventilation and breathlessness in outpatients with COPD. The study will not be blinded for participants and staff (due to the nature of the intervention) but will be blinded for the analyst.

The intervention is one night without sleep, and the control is one night with normal sleep. The test is a bicycle test (exercise test on a bike with continuous analysis of ventilation and gaseous exchange) carried out as a sub-max test at 75% of maximum capacity until the test person cannot go on.

The study consists of three visits. At the first visit, informed consent is collected, and inclusion and exclusion criteria are evaluated. Also, information is collected regarding the person's COPD-diagnosis, medication, and other illnesses. Specific surveys are Pittsburgh Sleep Quality Index (PSQI), COPD Assessment Test (CAT), modified Medical Research Council (mMRC) scale, 7-point Global Impression of Change (GIC) scale, Experienced sleep quality (Likert scale), Multidimensional Dyspnea Profile (MDP) to assess the person's sleep and respiration. Baseline values for dynamic spirometry, saturation, and blood pressure are also measured during the first visit. Afterwards, a bicycle test is carried out according to normal clinical standards. This involves increasing the resistance (in Watts) according to a set protocol until the test person is unable to continue. This takes roughly 6-10 minutes and provides a maximum performance value for the individual. This maximum value is used for visit number two and three. After this first visit the order of the sleepless night is randomized for either visit two or three.

At the second and third visit spirometry, saturation and blood pressure are once more measured. The person is evaluated for contraindications. Then a new bicycle test is carried out at 75% of the maximum W achieved at the first visit. The test takes around 10 minutes, and continues until the person is unable to continue. During this test, ventilation is measured as respiratory rate (RR), minute ventilation (MV), oxygen consumption (VO2), carbon dioxide consumption (VCO2), the respiratory quotient (VCO2/VO2), inspiratory capacity manoeuvre (IC), dynamic hyperinflation, ventilatory reserve capacity, ventilation efficiency (MV/VCO2-curve) and the anaerobic threshold. During the test the person is also assessed for how difficult the breathing feels (0-19 Borg CR10), how tired the legs feels (Borg CR10), how uncomfortable the breathing feels (mBorg 0-10) every two minutes and at the end of the test. At the end of the test the test person is asked about the reason for ending the test, how the breathing was experienced (Multidimensional Dyspnea Profile, MDP), and how motivated they were to carry out the test (0-10 NRS). The person is also monitored with EKG during the test, and the blood pressure is measured every two minutes. The results are then compared between the test where the person had a normal night's sleep, and the test where the person was awake the whole night before.

The normal night's sleep is assessed using some simple questions, such as: "How did you sleep tonight" and "How satisfied are you with the night's sleep?". It is also evaluated using an Actigraph bracelet that measures movement when worn. The bracelet is worn for 48 hours preceding both tests.

The night when the person is going to be awake is spent at the test lab, after eating a normal dinner at home. They then spend an entire night in a room where they can watch TV, use a phone or tablet or read books and magazines. They will be monitored by staff to help them stay awake during the night. They cannot eat, drink or smoke anything not usually consumed during the night (other than water). They then eat a normal breakfast of their choosing, and the test is carried out just like the one where they slept normally.

ELIGIBILITY:
Inclusion Criteria: (All required)

* Age 18 years or older
* COPD diagnosed by physician in accordance with Global Initiative For Chronic Obstructive Lung Disease (GOLD) guidelines (GOLD 2021), with a spirometric ratio of the forced expired volume in one second (FEV1) / forced vital capacity (FVC) < 0.7 and a FEV1 < 80% of predicted post bronchodilator at baseline.
* Self-reported average sleep time of six hours or longer during a normal night.
* No regular treatment with sleep medication or anxiolytics.
* Able to cycle
* Able to talk and write Swedish well enough to participate in the study procedures, as judged by the Investigator.

Exclusion Criteria:

* Resting peripheral oxygen saturation (SpO2) < 92%
* Night shift worker
* Hospitalization or clinical instability during the last four weeks
* Treatment with supplementary oxygen at rest or during exercise
* Sleep disturbance, defined as a Pittsburgh Sleep Quality Index >5 at baseline
* Contraindication to exercise testing in accordance with clinical practice guidelines (ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med 2003; 167:211-277)
* Expected survival shorter than six months as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in breathlessness intensity (Borg CR10) between control and intervention at iso-time | Measured during post-control and post-intervention exercise tests, spaced 7 days to 6 weeks apart
  Change between conditions in breathlessness intensity using the Borg Category Ratio scale (Borg CR10), where 0 indicates no exertion and 10 indicates maximum exertion, at iso-time (defined as the time of the latest similar time point during both conditions (control and intervention) during a constant rate cycle cardiopulmonary exercise test (CPET).

SECONDARY OUTCOMES:
Change in breathlessness unpleasantness (Borg CR10) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Perceived unpleasantness from breathlessness, measured with the Borg CR10 scale, where 0 indicates no exertion and 10 indicates maximum exertion. Compared at end exercise and at iso-time.
Change in time to the limit of tolerance (tLIM) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  For how long the test person can continue the test, measured in seconds.
Change in oxygen consumption between control and intervention (absolute) | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Measured using 7V'O2 (aerobic exercise capacity), in absolute numbers. Compared between the tests at peak exercise and at iso-time.
Change in oxygen consumption between control and intervention (%pred) | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Measured using V'O2, (aerobic exercise capacity), in percent of predicted (%pred). Compared between the tests at peak exercise and at iso-time.
Change in workload (W) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Maximum workload achieved, measured in Watts, in absolute numbers.
Change in workload (%pred) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Maximum workload achieved, measured in percent of predicted (%pred).
Change in Minute ventilation (VE) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Minute ventilation is measured and compared between the tests at peak exercise and at iso-time.
Change in tidal volume (VT) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Tidal volume measured and compared between the tests at peak exercise and at iso-time.
Change in ventilatory reserve, (MVV) - (VE) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Ventilatory reserve defined as maximum voluntary ventilation (MVV) - (VE). Compared between the tests at peak exercise and at iso-time.
Change in cardiac reserve between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Cardiac reserve is evaluated using the predicted peak heart rate. Compared between the tests at peak exercise and at iso-time.
Change in dynamic hyperinflation and inspiratory capacity (IC) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  This includes measures of constrained ventilatory expansion such as the inspiratory reserve volume (IRV). Compared between the tests at peak exercise and at iso-time.
Change in breathing frequency between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Breathing frequency is measured, and compared between the tests at peak exercise and at iso-time.
Change in breathlessness intensity at peak exercise (Borg CR10) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Perceived breathlessness intensity at peak exercise is evaluated using the Borg CR10 scale, where 0 indicates no exertion and 10 indicates maximum exertion, and compared between the tests.
Change in leg discomfort (Borg CR10) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Perceived leg discomfort is evaluated using the Borg CR10 scale, where 0 indicates no exertion and 10 indicates maximum exertion, and compared between the tests.
Change in timing of the anaerobic threshold (AT) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  At the anaerobic threshold, timing is registered, and compared between the tests.
Change in V'O2 of the anaerobic threshold (AT) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  At the anaerobic threshold, V'O2 is registered, and compared between the tests.
Change in efficacy of ventilation (VE/V'CO2-slope and ratio at the AT) between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  VE/V'CO2-slope and ratio are evaluated at the anaerobic threshold, and compared between the tests.
Change in respiratory exchange ratio (RER), defined as V'CO2/V'O2 between control and intervention | Measured during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Respiratory exchange ratio is calculated using V'CO2/V'O2, and compared between the tests at peak exercise and at iso-time.
Change in causes for stopping the test between control and intervention | Evaluated during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  The test person's reason for discontinuing the test is recorded.
Change in any adverse events during the control and intervention tests | Evaluated during post-control and post-intervention tests, spaced 7 days to 6 weeks apart
  Any adverse events during the tests are recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Blekinge Tekniska Högskola (BTH), Karlskrona, Blekinge County
  - Department of Clinical Physiology, Blekinge Hospital, Karlskrona, Blekinge County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Donnell DE, Banzett RB, Carrieri-Kohlman V, Casaburi R, Davenport PW, Gandevia SC, Gelb AF, Mahler DA, Webb KA. Pathophysiology of dyspnea in chronic obstructive pulmonary disease: a roundtable. Proc Am Thorac Soc. 2007 May;4(2):145-68. doi: 10.1513/pats.200611-159CC. PMID 17494725
- [Background] Agusti A, Edwards LD, Celli B, Macnee W, Calverley PM, Mullerova H, Lomas DA, Wouters E, Bakke P, Rennard S, Crim C, Miller BE, Coxson HO, Yates JC, Tal-Singer R, Vestbo J; ECLIPSE Investigators. Characteristics, stability and outcomes of the 2011 GOLD COPD groups in the ECLIPSE cohort. Eur Respir J. 2013 Sep;42(3):636-46. doi: 10.1183/09031936.00195212. Epub 2013 Jun 13. PMID 23766334
- [Background] Simon ST, Bausewein C, Schildmann E, Higginson IJ, Magnussen H, Scheve C, Ramsenthaler C. Episodic breathlessness in patients with advanced disease: a systematic review. J Pain Symptom Manage. 2013 Mar;45(3):561-78. doi: 10.1016/j.jpainsymman.2012.02.022. Epub 2012 Aug 24. PMID 22921180
- [Background] Dharmarajan K, Swami S, Gou RY, Jones RN, Inouye SK. Pathway from Delirium to Death: Potential In-Hospital Mediators of Excess Mortality. J Am Geriatr Soc. 2017 May;65(5):1026-1033. doi: 10.1111/jgs.14743. Epub 2016 Dec 30. PMID 28039852
- [Background] Rault C, Sangare A, Diaz V, Ragot S, Frat JP, Raux M, Similowski T, Robert R, Thille AW, Drouot X. Impact of Sleep Deprivation on Respiratory Motor Output and Endurance. A Physiological Study. Am J Respir Crit Care Med. 2020 Apr 15;201(8):976-983. doi: 10.1164/rccm.201904-0819OC. PMID 31810378
- [Background] Chen R, Tian JW, Zhou LQ, Chen X, Yan HY, Zeng B, Zhang MS. The relationship between sleep quality and functional exercise capacity in COPD. Clin Respir J. 2016 Jul;10(4):477-85. doi: 10.1111/crj.12249. Epub 2015 Jan 15. PMID 25515647
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Hedenstrom H, Malmberg P, Fridriksson HV. Reference values for lung function tests in men: regression equations with smoking variables. Ups J Med Sci. 1986;91(3):299-310. doi: 10.3109/03009738609178670. PMID 3811032
- See also: Related Info — https://goldcopd.org/wp-content/uploads/2020/11/GOLD-REPORT-2021-v1.1-25Nov20_WMV.pdf